CLINICAL TRIAL: NCT07137897
Title: Telerehabilitation of Patients With Osteoarthritis of the Knee Joint: Study Protocol for a Randomised Controlled Trial
Brief Title: Telerehabilitation for Knee Osteoarthritis: Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novo Mesto (Other)
Responsible Party: Principal Investigator, Karmen Erjavec, Principal Investigator, University of Novo Mesto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L7-50184
Record Dates: First submitted 2025-03-24; First posted 2025-08-22 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-03

CONDITIONS: Pain; Stiffness; Physical Function
Keywords: Telerehabilitation; knee; osteoarthritis; RCT; Physical Activity
MeSH Terms: conditions — Pain; Osteoarthritis; Motor Activity | interventions — Telerehabilitation; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): Patients in the Telerehabilitation group will receive instructions on physiotherapy intervention. They will independently perform the exercise for at least three months. During this time, they will have access to continuous remote support from the physiotherapist, including: • Weekly scheduled phone consultations • Live virtual consultations via MS Teams, Zoom, or Skype • Text messages and emails for personalised guidance, motivation, and ongoing problem solving.
  Interventions: Other: Control group
- Control group (Active Comparator): Patients in the control group will receive only written exercise instructions and perform the rehabilitation program independently at home without additional remote supervision.
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Telerehabilitation involves a physiotherapy program delivered remotely using digital tools. Participants perform exercises independently with remote support from a physiotherapist, including:
  Weekly scheduled phone consultations
  Live virtual consultations via MS Teams, Zoom, or Skype
  Text messages and emails for personalized guidance, motivation, and ongoing problem-solving
  The intervention includes targeted exercises for:
  Core muscle strength
  Strengthening of lower extremity muscles
  Mobility exercises for the hip, knee, and ankle joints
  Balance and stabilization exercises
  Each session lasts approximately 20-25 minutes, performed three times per week. Patients can choose the days for their sessions, with the requirement of a minimum of 24 hours and a maximum of 72 hours of rest between sessions.
  The intervention will last for at least three months.
  Arms: Control group
Other: Control group — Patients in the control group will receive written instructions for a home exercise program. They will independently perform the rehabilitation program at home without remote supervision.
  The intervention includes targeted exercises for:
  Core muscle strength
  Strengthening of lower extremity muscles
  Mobility exercises for the hip, knee, and ankle joints
  Balance and stabilization exercises
  Each session lasts approximately 20-25 minutes, performed three times per week. Patients can choose the days for their sessions, with the requirement of a minimum of 24 hours and a maximum of 72 hours of rest between sessions.
  The intervention will last for at least three months.
  Arms: Telerehabilitation Group

SUMMARY:
Patient Recruitment and Enrolment

All patients diagnosed with knee OA who present at Artros Medical Center for an orthopaedic specialist consultation will undergo a radiological examination. Based on the radiographic findings and clinical evaluation, the orthopaedic specialist will refer eligible patients to a physiotherapist, who will assign them to the TG or CG. The physiotherapist will provide both verbal and written explanations of the study procedures. Patients will be included in the study after providing written informed consent.

Baseline Assessments

The physiotherapist will collect baseline data, including: Sociodemographic characteristics, Anthropometric measurements: height (cm), weight (kg), body mass index (BMI) (kg/m²), Educational background and employment status, Knee joint mobility assessment using a goniometer, Pain intensity measurement using the Numerical Rating Scale (NRS), Physical function, stiffness, and pain assessment using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Physical activity evaluation using the International Physical Activity Questionnaire (IPAQ), Health-related quality of life assessment using the 12-Item Short Form Health Survey (SF-12), OA severity classification based on recent knee radiographs (≤ 4 months old), graded using the Kellgren-Lawrence classification system.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee is a chronic degenerative disease that affects the articular cartilage, causing pain, reduced mobility and reduced quality of life. Early detection and appropriate treatment are key to reducing symptoms and slowing disease progression. This study aims to evaluate the effectiveness of therapeutic interventions in patients with knee OA treated at the Artros Medical Centre.

Patients diagnosed with OA of the knee who visit the Artros Medical Centre for a consultation with an orthopaedic specialist will be included in the study. After the visit, they will undergo a radiological examination, based on which the orthopaedic surgeon will assess the severity of the disease. The specialist will then refer suitable patients to a physiotherapist who will further assess them and assign them to a telerehabilitation group (TR) or a control group (TS). The physiotherapist will provide verbal and written explanations of the study procedures to the patients.

Written informed consent will be required from each participant to participate in the study.

After inclusion in the study, the physiotherapist will collect baseline data on the patients, including the following measures:

* Sociodemographic characteristics: age, gender, education, employment status.
* Anthropometric measurements: height (cm), weight (kg), body mass index (BMI) (kg/m²).
* Assessment of knee joint mobility: measurement of range of movement with a goniometer.
* Pain intensity: Use the Numerical Rating Scale (NRS) to measure subjective pain.

Assessment of physical function, stiffness, and pain: The validated Western Ontario and McMaster University Osteoarthritis Index (WOMAC) questionnaire is used.

* Physical activity assessment: performed using the International Physical Activity Questionnaire (IPAQ).
* Assessment of health-related quality of life: administered by the 12-item Short Form Health Survey (SF-12).
* Osteoarthritis severity classification: based on knee radiographs (≤ 4 months old) and will be performed according to the Kellgren-Lawrence classification system.

Patients will be randomly assigned to one of two groups:

* telerehabilitation group (TR): They will be enrolled in a tailored physiotherapy programme, including individually tailored exercises to strengthen, stretch, and improve the functionality of the knee joint.
* control group (CG): patients will continue with standard care without additional therapeutic interventions.

Patient measurements and assessments will be carried out at the start of the study and at specific time points (after 12 weeks). All data will be recorded and analysed to identify changes in pain, mobility, functionality, and quality of life.

Statistical analysis Data will be analysed using appropriate statistical methods (e.g., t-test, ANOVA, regression analysis). The main outcome parameters will be changes in WOMAC, NRS, IPAQ, and SF-12, where the statistical significance and clinical relevance of differences between groups will be assessed.

The Declaration of Helsinki will conduct the study, which will be subject to ethics committee approval. Before participation, all participants will be informed in detail about the nature of the study and the potential risks and benefits, and their inclusion will be voluntary.

This study will provide valuable data on the effectiveness of therapeutic interventions in patients with knee OA and will contribute to a better understanding of optimal approaches to treating this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic OA of the knee joint, graded 1-3 on the Kellgren-Lawrence scale
2. Patients older than 50 years
3. Patients with access to and proficiency in using a computer,
4. Patients with the capability to follow the exercises outlined.

Exclusion Criteria:

1. Grade 4 cartilage defect (cartilage defect up to the subchondral bone), for which surgical treatment is professionally indicated,
2. Planned arthroplasty of the knee joint within the next 6 months,
3. Patients who have had a previous TEP arthroplasty or partial knee arthroplasty (hereafter PEP),
4. Patients with a history of trauma or surgical treatment of the knee joint (osteotomy or treatment of cartilage lesions) in the last 6 months,
5. Patients who have received an intra-articular injection in the knee joint in the last 3 months,
6. Patients who have systemic inflammatory arthritis (e.g. rheumatoid arthritis or gout) or those who have concomitant medical conditions that prevent participation in exercise,
7. Patients who have cognitive impairments or are wheelchair users,
8. Who has co-morbidities,
9. Those who do not have access to a computer have limited language skills that prevent the correct use of tele-rehabilitation or
10. Those who are involved in similar study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Day 1
  Measured using the Numeric Rating Scale (NRS), where the scale ranges from 0 to 10, with 0 representing 'no pain' and 10 representing 'worst possible pain'. Higher scores indicate a higher level of pain.
Knee Function (WOMAC) | Day 1
  Evaluated using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), which measures joint function, stiffness, and pain related explicitly to knee osteoarthritis.
Joint Mobility | Day 1
  Joint mobility will be assessed using a goniometer to measure any improvements or changes in the range of motion of the knee joint.
Physical Activity | Day 1
  Assessed using the International Physical Activity Questionnaire (IPAQ), gauges the level of physical activity and sedentary behaviour in daily life. Health-Related
Quality of Life ( SF-12) | Day 1
  Measured by the SF-12, a 12-item questionnaire that evaluates the patient's perceived quality of life, focusing on physical and mental health.

SECONDARY OUTCOMES:
Pain Intensity | up to 12 weeks
  Measured using the Numeric Rating Scale (NRS) to assess changes in pain levels experienced by patients during rehabilitation and following the intervention.
Knee Function (WOMAC) | up to 12 weeks
  Evaluated using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), which measures joint function, stiffness, and pain related explicitly to knee osteoarthritis.
Physical Activity | up to 12 weeks
  Assessed using the International Physical Activity Questionnaire (IPAQ), gauges the level of physical activity and sedentary behaviour in daily life.
Quality of Life ( SF-12) | up to 12 weeks
  Measured by the SF-12, a 12-item questionnaire that evaluates the patient's perceived quality of life, focusing on physical and mental health.
Exercise Adherence and Frequency | up to 12 weeks
  Monitoring the regularity and consistency with which patients in both TG and CG complete the prescribed exercises, along with any challenges encountered that may influence adherence.
Patient Satisfaction with telerehabilitation | up to 12 weeks
  Following the intervention, patients will provide feedback on their overall satisfaction with the telerehabilitation approach, including perceived benefits and limitations.
Reasons for Reduced Exercise Engagement or Discontinuation | up to 12 weeks
  Patients will report any factors contributing to decreased exercise frequency or halting the rehabilitation program, particularly in the TG.
Joint Mobility | up to 12 weeks
  Joint mobility will be reassessed using a goniometer to measure any improvements or changes in the range of motion of the knee joint.

CONTACTS AND LOCATIONS:
Overall Officials: Karmen Erjavec, prof. dr., Study Director — University of Novo Mesto
Locations (1):
- University of Novo mesto Faculty of Health Sciences, Novo Mesto, Slovenia